CLINICAL TRIAL: NCT06095622
Title: Formulation and Assessment of Chickpea Pulao Using Fenugreek Seeds and Indian Rennet for Improving Blood Glycemic Levels
Brief Title: Chickpea Pulao Using Fenugreek Seeds and Indian Rennet for Improving Blood Glycaemic Levels
Acronym: DP-Trails
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Management and Technology Lahore (Other)
Responsible Party: Principal Investigator, Nauman Khalid, Professor, University of Management and Technology Lahore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022-03-R002-C-1
Record Dates: First submitted 2023-10-01; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus)
Keywords: Chickpea pulao; Fenugreek seeds; Indian rennet; Glucose modulating
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Typical rice pulao without and herbal intervention (No Intervention): Normal chickpea rice pulao was used as the main arm. The control group does not contain fenugreek and Indian rennet extract.
- Chickpea Pulao Using Fenugreek Seeds and Indian Rennet (Experimental): Chickpea rice pulao added with herb (Fenugreek Seeds and Indian Rennet).
  Interventions: Dietary Supplement: Fenugreek Seeds and Indian Rennet

INTERVENTIONS:
Dietary Supplement: Fenugreek Seeds and Indian Rennet — Food herbs like fenugreek Seeds and Indian rennet to formulate rice dish.
  Arms: Chickpea Pulao Using Fenugreek Seeds and Indian Rennet

SUMMARY:
The goal of this study was to perform a clinical trial to compare the impact of herbal chickpea pulao (cooked Indian-Pakistani rice dish) on improving postprandial blood glucose levels in type-2 diabetic people. The main questions it aims to answer are:

* Whether Indian rennet and fenugreek seed extract can modulate blood sugar levels or not?
* At what concentration the flavor, taste, and blood sugar impact were acceptable?

Participants were provided with control and intervention herbal chickpea pulao for a period of 21 days and asked to provide feedback on taste, flavor, and over-acceptability, and their postprandial blood glucose levels were checked.

ELIGIBILITY:
Inclusion Criteria:

* People having Type-2 diabetes disease
* Must be able to consume chickpea rice pulao
* Must not be on vegan or keto diet

Exclusion Criteria:

* Healthy people without diabetes
* People with less than 18 years of age

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Improvement in blood glucose levels | 21 days
  Increase or decrease in postprandial glucose levels in mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Management and Technology, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The results data collected, de-identified individual participant data, and composition of recipe will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after the publication of the manuscript.
Access Criteria: The data can be requested from the corresponding author.